CLINICAL TRIAL: NCT01448187
Title: Descriptive Pharmacoepidemiological Study of Patients Treated With Iressa
Acronym: EPIDAURE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-OFR-IRE-2011/1
Record Dates: First submitted 2011-09-26; First posted 2011-10-07 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-07

CONDITIONS: Lung Cancer
Keywords: Lung cancer, France
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the study is to describe the characteristics of patients treated with Iressa (particularly age, gender, phenotype, histology and stage of disease, line of treatment and previous treatments, smoking history, conditions of initiation of treatment (presence of an EGFR-activating mutation) and to evaluate the impact of treatment on the health of the population concerned in terms of morbidity and mortality (clinical benefit, safety,...) and quality of life

DETAILED DESCRIPTION:
Descriptive pharmacoepidemiological study of patients treated with Iressa

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with Iressa

Exclusion Criteria:

* Patient included in a therapeutic trial comprising protocol use of Iressa
* Patient included in a therapeutic trial (Huriet-Serusclat Act)
* Patient refusing to participate in the study

Max Age: 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospital, clinic
Sampling Method: Probability Sample
Enrollment: 361 (Actual)
Dates: Start 2012-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
The Overall survival | 24 months
The progression free survival | 24 months

SECONDARY OUTCOMES:
Description of Quality of life by Functional Assessment of Cancer Therapy - Lung including Life Stressor Checklist (FACT-L including LSC) | baseline
Description of Quality of life by Functional Assessment of Cancer Therapy - Lung including Life Stressor Checklist (FACT-L including LSC) | From baseline to 3 months
Description of Quality of life by Life Stressor Checklist - Lung (LSC-L) | From 3 months to 6 months
Description of Quality of life by Life Stressor Checklist - Lung (LSC-L) | From 6 months to 12 months
Description of Quality of life by Life Stressor Checklist - Lung (LSC-L) | From 12 months to 18 months
Description of Quality of life by Life Stressor Checklist - Lung (LSC-L) | From 18 months to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Thierry BOUILLET, Dr, Principal Investigator — Bobigny; Elisabeth BRAMBILLA, Pr, Principal Investigator — Grenoble; Jacques CADRANEL, Pr, Principal Investigator — Paris; Jean-Francois MORERE, Pr, Principal Investigator — Bobigny; Maurice PEROL, Dr, Principal Investigator — Lyon; Virginie RONDEAU, PhD, Principal Investigator — Bordeaux
Locations (29):
- France (29):
  - Research Site, Aulnay-sous-Bois
  - Research Site, Bayonne
  - Research Site, Bordeaux
  - Research Site, Bron
  - Research Site, Carcassonne
  - Research Site, Chalon-sur-Saône
  - Research Site, Cholet
  - Research Site, Clamart
  - Research Site, Colmar
  - Research Site, Corbeil-Essonnes
  - Research Site, Créteil
  - Research Site, Épernay
  - Research Site, La Source
  - Research Site, Marseille
  - Research Site, Mâcon
  - Reseacrh Site, Metz
  - Research Site, Mont-de-Marsan
  - Research Site, Niort
  - Research Site, Paris
  - Research Site, Pierre-Bénite
  - Research Site, Quimper
  - Research Site, Reims
  - Research Site, Rouen
  - Research Site, Saint-Herblain
  - Research Site, Saint-Nazaire
  - Research Site, Saint-Omer
  - Research Site, Strasbourg
  - Research Site, Toulon
  - Research Site, Vienne

REFERENCES:
- See also: NIS-OFR-IRE-2011_1CSR_Synopsis.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=995&filename=NIS-OFR-IRE-2011_1_CSR_Synopsis%20.pdf